CLINICAL TRIAL: NCT05920187
Title: Additive Modified Mediterranean Dietary Intervention Versus Modified Anti-inflammatory Dietary Intervention for Inflammatory Bowel Disease Remission
Brief Title: Dietary Intervention for Inflammatory Bowel Disease Remission
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Khaled Mostafa Mohamed, Assistant lecturer of Tropical Medicine and Gastroenterology, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: dietary intervention in IBD
Record Dates: First submitted 2023-03-18; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Diet, Mediterranean; Insemination, Artificial, Heterologous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mediterranean diet group (Active Comparator): following dietary intervention based on Mediterranean diet
  Interventions: Other: Mediterranean diet and Anti-inflammatory diet
- Anti-inflammatory diet group (Active Comparator): following dietary intervention based on IBD-Anti-inflammatory diet.
  Interventions: Other: Mediterranean diet and Anti-inflammatory diet
- control group (No Intervention): Patients of the control group will not be instructed to follow a specific dietary intervention.

INTERVENTIONS:
Other: Mediterranean diet and Anti-inflammatory diet — Cases will be randomly allocated to two groups: Mediterranean diet group (following dietary intervention based on MD), and Anti_inflammatory diet group(following dietary intervention based on IBD-AIF). Patients of the control group will not be instructed to follow a specific dietary intervention.
  Evaluation of adherence of cases to dietary intervention will be at two points of time: after four weeks and after 12 weeks by using Mediterranean Diet Serving Score (MDSS) for MD adherence and Anti- Inflammatory Diet Serving Score for IBD- AID adherence. The AID Serving Score (AIDSS) is based on the latest update of the Anti-Inflammatory Diet Pyramid, using the recommended consumption frequency of foods and food group.
  Other Names: MD and AID
  Arms: Anti-inflammatory diet group; Mediterranean diet group

SUMMARY:
1. To compare adding dietary intervention based on MD to dietary intervention based on IBD-AID on induction of disease remission of IBD patients receiving pharmacotherapy.
2. To compare patients' adherence to dietary intervention based on MD to dietary intervention based on IBD-AID, and the impact of adherence on induction of remission among patients with IBD receiving pharmacotherapy.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic inflammatory disorder with two major types; ulcerative colitis (UC) and Crohn's disease (CD) . There is a growing incidence of IBD in the Arab world, with incidence rate of 2.33 per 100,000 persons per year for UC and 1.46 per 100,000 persons per year for CD.

Due to this increasing incidence, it is likely that IBD will become a major health problem in the future.

Pathogenesis of IBD is not fully understood yet, recent studies suggest that IBD is associated with a multifactorial process involving genetics, environmental factors, microbiota, and deregulation of the immune system.

Diet is one of the environmental factors involved in the onset and course of IBD. Accumulating evidence points to gut dysbiosis combined with aberrant immune response in genetically predisposed individuals; a process probably triggered and maintained by changes in environmental factors, including diet ; the exact interplay between these factors is still unknown.

Since the prevalence of IBD is highest in the Western world, affecting up to 0.5% of the general population in 2015, it is thought that the Western diet, high in fats and sugars and low in vegetables and fruits, contributes to the development of IBD.

Several diets have been proposed for the treatment or prevention of different diseases. One of the most widely used is the Mediterranean diet (MD), which was recently suggested for management of several diseases. The traditional Mediterranean diet is characterized by high consumption of vegetables, fruits, olive oil, nuts, and legumes, as well as fish and unprocessed cereals, low intake of meat, meat products, and dairy products .

Another diet, the IBD anti-inflammatory diet (AID) which restricts intake of certain carbohydrates and includes pre- and probiotic foods and modified dietary fatty acids showed some improvements in a case series study as adjunct dietary therapy for treatment of IBD patient.

Application of healthier dietary patterns has been considered effective, non-invasive, and long-lasting therapy. Therapeutic diets should be evaluated as an adjunct therapy to reduce number and/or dose of IBD medications, with consequent reduction of cost and adverse effects. However, high-quality data to guide the dietary recommendations are still lacking.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of IBD (according to clinical, endoscopic and histological criteria).

  * Receiving pharmacotherapy for IBD.

Exclusion Criteria:

* Pediatric patients (less than 18 years old)
* Pregnant or breastfeeding patients
* Patients with concomitant alimentary tract disorders, such as malabsorption and celiac disease
* Patients requiring specific dietary interventions, such as diabetes mellitus, heart failure, renal failure, nephrosis, and liver failure, and neoplastic disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Induction of disease remission by adding adjunct dietary interventions combined with pharmacotherapy. | 12 weeks
  by standard biochemical procedures, such as C-reactive protein (CRP).
Induction of disease remission by adding adjunct dietary interventions combined with pharmacotherapy. | 12 weeks
  standard biochemical procedures, such as C-reactive protein (CRP) and fecal calprotectin (FC) levels.
Induction of disease remission (UC) by adding adjunct dietary interventions combined with pharmacotherapy. | 12 weeks
  For UC patients, Clinician based Simple Clinical Colitis Activity Index (SCCAI) categorize two types of patients: patients with inactive disease (SCCAI score < 5) and patients with active disease (SCCAI score ≥ 5).
Induction of disease remission (UC) by adding adjunct dietary interventions combined with pharmacotherapy. | 12 weeks
  by using Mayo score/disease activity index (Mayo/DAI) A score of 3 to 5 points indicates mildly active disease, a score of 6 to 10 points indicates moderately active disease, and a score of 11 to 12 points indicates severely active disease.
Induction of disease remission (CD) by adding adjunct dietary interventions combined with pharmacotherapy. | 12 weeks
  . For Crohn's disease patients, Modified Harvey Bradshaw Index will be used with score ≤ 5 indicate remission, =5-7mild disease ,8-16 moderate disease, ≥ 16 in severe disease.

SECONDARY OUTCOMES:
Adherence of IBD patients to adjunct dietary interventions, and its impact on induction of remission. | 12 Weeks
  will be at two points of time: after four weeks and after 12 weeks by using Mediterranean Diet Serving Score (MDSS) (16) for MD adherence.
Adherence of IBD patients to adjunct dietary interventions, and its impact on induction of remission. | 12 weeks
  will be at two points of time: after four weeks and after 12 weeks by using Anti- Inflammatory Diet Serving Score for IBD- AID adherence. The AID Serving Score (AIDSS) is based on the latest update of the Anti-Inflammatory Diet Pyramid, using the recommended consumption frequency of foods and food group.

IPD SHARING:
Plan to Share IPD: Yes